CLINICAL TRIAL: NCT00139841
Title: A Multi-Center Phase III Study to Investigate the Safety and Efficacy of Treanda™ (Bendamustine HCl) in Patients With Indolent Non-Hodgkin's Lymphoma (NHL) Who Are Refractory to Rituximab
Brief Title: Safety and Efficacy of Treanda™ (Bendamustine HCl) in Patients With Indolent Non-Hodgkin's Lymphoma (NHL) Who Are Refractory to Rituximab
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cephalon (Industry)
Responsible Party: Sponsor
Organization: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SDX-105-03
Record Dates: First submitted 2005-08-18; First posted 2005-08-31 (Estimated); Last update posted 2014-05-09 (Estimated); Status verified 2014-05

CONDITIONS: Non-Hodgkin's Lymphoma
Keywords: Lymphoma, Non-Hodgkin; Rituximab Refractory; Rituximab Failure; Indolent Non-Hodgkins Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — Bendamustine Hydrochloride

ARMS (1):
- 1 (Experimental): bendamustine
  Interventions: Drug: Bendamustine HCl

INTERVENTIONS:
Drug: Bendamustine HCl — Dose of 120 mg/m2 on Day 1 and Day 2 of each treatment cycle (every 21 days). Patients who are continuing to experience clinical benefit at Cycle 6, as assessed by the investigator, may receive up to 2 additional cycles, to a maximum of 8 cycles.

SUMMARY:
SUMMARY: This is a multi-center open label study to evaluate the safety and effectiveness of Treanda™ (also known as bendamustine HCl or SDX-105) in patients who have indolent Non-Hodgkin's lymphoma and have relapsed within a defined timeframe after taking rituximab (Rituxan®). Treanda will be given via 60-minute intravenous infusion on days 1 and 2 of every 21-day treatment cycle. Patients will be treated for 6 cycles unless they develop progressive disease or unacceptable toxicity. Those who continue to receive clinical benefit at end of 6 cycles may receive an additional 2 cycles. Following the end of treatment, patients will be followed for up to 2 years until disease progression or start of another anti-cancer therapy.

ELIGIBILITY:
ELIGIBILITY:

Key Inclusion Criteria

* Documented B-cell Non-Hodgkin's Lymphoma
* Small lymphocytic lymphoma (ALC < 5,000 cells/mm3)
* Marginal zone B-cell lymphoma (nodal, extranodal, or splenic types)
* Lymphoplasmacytic lymphoma
* Follicular center lymphoma, follicular

Disease documented to be refractory to a full-course of the most recent rituximab therapy (single agent or combination)

* At least 1 prior chemotherapy regimen and maximum of 3 prior chemotherapy regimens
* Bidimensionally measurable disease (by CT scan) with at least one lesion measuring ≥ 2.0 cm in a single dimension

Key Exclusion Criteria

* Patients who receive rituximab only as part of treatment with ibritumomab tiuxetan (Zevalin®) will not be eligible
* History of prior high dose chemotherapy with allogeneic stem cell support (history of autologous stem cell support is permissible)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2005-10; Primary Completion 2007-07 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Assess the overall response rate (ORR = CR + CRu + PR) and duration of response (DR) to a regimen of bendamustine in patients who are refractory to rituximab therapy. | 6 months

SECONDARY OUTCOMES:
• assess the safety profile of Treanda in this patient population. • assess the duration of progression-free survival (PFS). • estimate the basic pharmacokinetic parameters • assess the effects of plasma concentrations | 6 months

CONTACTS AND LOCATIONS:
Locations (40):
- United States (32):
  - University of Alabama Birmingham, Birmingham, Alabama
  - Arizona Cancer Center, Tucson, Arizona
  - Alta Bates Comprehensive Cancer Center, Berkeley, California
  - Tower Hematology and Oncology Medical Group, Beverly Hills, California
  - Moores UCSD Cancer Center, La Jolla, California
  - USC/Norris Cancer Hospital, Los Angeles, California
  - Comprehensive Cancer Center - Desert Regional Medical Center, Palm Springs, California
  - Stanford University Division of Oncology, Stanford, California
  - University of Colorado Cancer Center, Aurora, Colorado
  - Yale University School of Medicine, New Haven, Connecticut
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - Rush University Medical Center, Chicago, Illinois
  - Indiana Oncology Hematology Consultants, A Division of AHN, Indianapolis, Indiana
  - Markey Cancer Center, University of Kentucky Medical Center, Lexington, Kentucky
  - LSU Health Sciences Center, Feist Weiller Cancer Center, Shreveport, Louisiana
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan Cancer Center, Ann Arbor, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - Washington University School of Medicine in St. Louis, St Louis, Missouri
  - Nevada Cancer Institute, Las Vegas, Nevada
  - University of New Mexico Cancer Research and Treatment Center, Albuquerque, New Mexico
  - Roswell Park Cancer Institute, Buffalo, New York
  - Weill Cornell Cancer Care Center, New York, New York
  - Interlakes Foundation, Inc., Rochester, New York
  - University of Rochester Medical Center, James P. Wilmot Cancer Center, Rochester, New York
  - Duke University School of Medicine, Durham, North Carolina
  - The Cleveland Clinic Foundation Taussig Cancer Center, Cleveland, Ohio
  - The West Clinic/ACORN, Memphis, Tennessee
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Arlington Cancer Center, Arlington, Texas
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - University of Wisconsin, Madison, Wisconsin
- Canada (7):
  - Cross Cancer Institute, Edmonton, Alberta
  - British Columbia Cancer Agency, Vancouver, British Columbia
  - Queen Elizabeth Health Sciences Centre, Halifax, Nova Scotia
  - Ottawa Hospital - General Campus, Ottawa, Ontario
  - Hopital Notre-Dame du CHUM, Montreal, Quebec
  - Hopital du Sacre Couer de Montreal, Montreal, Quebec
  - Saskatchewan Cancer Center Agency, Saskatoon, Saskatchewan
- Hospital Espanol Auxilio Mutuo, Auxilio Mutuo Cancer Center, San Juan, Puerto Rico